CLINICAL TRIAL: NCT01409967
Title: The Impact of Red Packed Cells Transfusion on the Main Biological Markers to Determine the Etiology of Anemias
Acronym: BÉA/T
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10060; HAO 10048 (Other: Management number)
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Anemia
Keywords: Anemia; Transfusion; Biological markers
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this work is to study the changes of key assays useful for the understanding of anemia mechanism before and after red packed cells transfusion: iron status, vitamin assays, hemolysis markers.

DETAILED DESCRIPTION:
The aim of this work is to study the changes of key assays useful for the understanding of anemia mechanism before and after red packed cells transfusion: iron status, vitamin assays, hemolysis markers.

The patient selection criteria are:

* age > or = 18 years
* No history of transfusion > or = 2 years
* Anemia (any etiology known or assumed)
* Decision of red packed cells transfusion for the current episode
* Transfusion performed at BEAUJON Hospital
* Agreement of patient for the study

Number of subjects required: 100 patients

Study duration and duration of participation for each patient:

* duration of the study: 1 year
* for each patient the participation to the study began at baseline after the decision of transfusion and stopped at the second sample ie at least 72 hours after the transfusion of red blood cells.

The maximum contribution for one patient is 5 days.

Methodology: It is a prospective non interventional monocentric (BEAUJON Hospital) study. Two blood tests will be performed; one before transfusion and the other from 48 to 72 hours after red packed cells transfusion.

The following parameters will be measured before and after red packed cells transfusion:

Complete blood count (CBC) with reticulocyte count; complete iron status (ferritin, serum iron, transferrin, transferrin saturation), soluble transferrin receptor; serum and intraerythrocytic folate levels, vitamin B12; lactate dehydrogenase (LDH), bilirubin (total and free), haptoglobin, orosomucoid, direct coombs test; creatinine; CRP.

The aim of this work is to study the changes of key assays useful for the understanding of anemia mechanism before and after red packed cells transfusion: iron status, vitamin assays, hemolysis markers.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age > or = 18 years
* No history of transfusion > or = 2 years
* Anemia (any etiology known or assumed)
* Decision of red packed cells transfusion for the current episode
* Transfusion performed at BEAUJON Hospital
* Agreement of patient for the study

EXCLUSION CRITERIA:

* Patient who received between the 2 samples, a treatment which can modify the parameters evaluated (iron, vitamin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemic patient with decision of red packed cells transfusion for the current episode.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
anemia | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Froissart Antoine, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital BEAUJON, Clichy, France